CLINICAL TRIAL: NCT01750268
Title: Topiramate Treatment of Hazardous and Harmful Alcohol Use in Veterans With TBI
Acronym: VAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Northern California Institute of Research and Education (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-11-2-0145
Record Dates: First submitted 2012-11-28; First posted 2012-12-17 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury (TBI); Hazardous and Harmful Alcohol Use
Keywords: TBI; hazardous and harmful alcohol use; veterans; co-occurring disorders; pharmacotherapy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): Topiramate capsules daily - up to 300 mg
  Interventions: Behavioral: Medical Management Counseling; Drug: Topiramate
- Placebo (Placebo Comparator): Placebo capsules daily - up 300 mg
  Interventions: Behavioral: Medical Management Counseling; Drug: Placebo

INTERVENTIONS:
Behavioral: Medical Management Counseling — Brief alcohol and medication counseling
Drug: Topiramate — Experimental medication
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The goal of the proposed project is to improve the treatment of veterans with co-occurring traumatic brain injury (TBI) and hazardous or harmful alcohol use. The PI and coinvestigators will conduct a pilot controlled clinical trial of topiramate for the treatment of these co-occurring disorders.

ELIGIBILITY:
Inclusion Criteria

1. Male and female veterans.
2. Ages 18 to 65 (inclusive).
3. TBI: a history of mild traumatic brain injury, as defined by American Congress of Rehabilitation Medicine (ACRM) and VA, in the chronic, stable phase of recovery (>6 months from injury). The ACRM defines mild TBI as a traumatically-induced physiological disruption of brain function as demonstrated by at least one of the following:

3.a. loss of consciousness of up to 30 minutes;

3.b. any loss of memory for events immediately before or after the event;

3.c. any alteration in mental state at the time of the event, for example feeling dazed, disoriented, or confused; and

3.d. a focal neurological deficit or deficits that may or may not have been transient, for example loss of coordination, speech difficulties, or double vision. ACRM's definition further specifies that a person may be designated as having a mild TBI only if the severity of the injury does not include a loss of consciousness that lasted longer than 30 minutes, and post-traumatic amnesia lasting longer than 24 hours.

Rationale:

1. This is the most common description of patients currently served by our VA facilities.
2. Studies at this stable phase will facilitate detection of otherwise subtle changes as findings are less likely to be confounded by 'spontaneous' recovery.

4. Current (past month) hazardous alcohol use or harmful alcohol use.

4.a. Hazardous use is drinking that must meet criteria for "at-risk" or "heavy" drinking by National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria: Subjects must report current (past 30 day) "at-risk" or "heavy" drinking on an average weekly basis, consisting of an average of 15 or more standard drinks per week for men and 8 or more standard drinks per week for women during the 30 days prior to Screening Visit 1 as measured by the Alcohol Timeline Followback (TLFB) method.

4.b. Harmful use is drinking behavior that meets Diagnostic and Statistical Manual (DSM)-IV diagnostic criteria for an Alcohol Use Disorder (Alcohol Dependence or Alcohol Abuse).

5. Subjects must express a desire to reduce or stop alcohol use.

6. Female subjects must have a negative urine pregnancy test and must be either postmenopausal for at least 1 year or practicing an effective method of birth control (e.g., surgically sterile, spermicide with barrier, male partner sterilization; or absent and agrees to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence).

7. Subjects must have a Breath Alcohol Concentration (BAC) of less than 0.02% when signing the informed consent form.

Exclusion Criteria

1. Psychotic disorders, bipolar disorders, dementia, or other psychiatric disorders judged to be unstable.
2. Subjects known to have clinically significant unstable medical conditions, including but not limited to: Clinically significant renal disease and/or impaired renal function as defined by clinically significant elevation of blood urea nitrogen (BUN) or creatinine or an estimated creatinine clearance of < 60 mL/min; AST and/or ALT > 5 times the upper limit of the normal range and/or a serum bilirubin > 2 times the upper limit of normal.
3. History of glaucoma.
4. History of kidney stones.
5. Concurrent participation in another alcohol treatment study or any study involving medications.
6. Female patients who are pregnant or lactating.
7. Topiramate use in the past week prior to study entry.
8. Use of medications for alcohol dependence (disulfiram, naltrexone, or acamprosate) within the past week.
9. Needing acute medical detoxification from alcohol based on a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD).
10. Subjects who are legally mandated to participate in an alcohol treatment program.
11. Subjects who have had a suicide attempt in the past 6 months or suicidal ideation, with intent, in the 30 days prior to enrollment.
12. Subjects who have previously been treated with topiramate for any reason and discontinued treatment due to an adverse event or due to a hypersensitivity reaction to topiramate.
13. Subjects with seizure disorders.
14. Subjects currently being treated with another anticonvulsant.
15. Subjects who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings or contraindications outlined in the topiramate package insert.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Batki, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Result] Pennington DL, Bielenberg J, Lasher B, Herbst E, Abrams G, Novakovic-Agopian T, Batki SL. A randomized pilot trial of topiramate for alcohol use disorder in veterans with traumatic brain injury: Effects on alcohol use, cognition, and post-concussive symptoms. Drug Alcohol Depend. 2020 Sep 1;214:108149. doi: 10.1016/j.drugalcdep.2020.108149. Epub 2020 Jul 2. PMID 32712569

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 15 | 17
Completed | 13 | 12
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (13.5) | 48.5 (14.0) | 46.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 10 | 15 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 4 | 9
  White | 7 | 9 | 16
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Drinking Days Per Week as Assessed by the Timeline Followback (TLFB)
Description: Using a calendar, participants provide retrospective estimates of daily drinking over a specified period.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Drinking Days per week
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 15 | 17
Drinking Days per week | 2.2 (1.8) | 1.6 (2.1)

2. Secondary Outcome: Change in TBI Symptom Severity as Assessed by the Neurobehavioral Symptom Inventory (NSI)
Description: Participants indicate the extent to which each of the 22 symptoms has disturbed them in the previous 2 weeks on a 5-item scale (0-none to 4-severe). The NSI total score is the sum of severity ratings of the symptoms. The scores are summed to yield a total score ranging from 0 to 88, where the higher the point value, the greater (more severe) the symptoms.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 15 | 17
scores on a scale | 16.3 (13.1) | 19.3 (15.1)

3. Other Pre Specified Outcome: Change in Alcohol Use as Assessed by the Timeline Followback (TLFB)
Description: Using a calendar, participants provide retrospective estimates of daily drinking over a specified period.
Time Frame: Baseline to Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, an average of 12 weeks
Arm/Group | Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 3/15 | 1/17
Other Adverse Events (participants affected / at risk) | 15/15 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=15) | Placebo (N=17)
Inpatient medical hospitalization for an episode of chest pain in the context of cocaine use (Cardiac disorders) | 1 (2) | 0 (0)
Voluntary psych inpatient admission due to homicidal ideation in the context of heavy cocaine use (Psychiatric disorders) | 1 (1) | 0 (0)
Inpatient medical hospitalization due to alcohol withdrawal (Psychiatric disorders) | 1 (1) | 0 (0)
Inpatient medical hospitalization for planned distal pancreatectomy and splenectomy (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=15) | Placebo (N=17)
Numbness and tingling (Nervous system disorders) | 5 | 5
Change in sense of taste (Nervous system disorders) | 8 | 5
Fatigue (General disorders) | 2 | 4
Loss of appetite (Gastrointestinal disorders) | 4 | 6
Difficulty with concentration and attention (Nervous system disorders) | 1 | 2
Nervousness (Psychiatric disorders) | 2 | 2
Difficulty with memory (Nervous system disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 3
Dizziness (Ear and labyrinth disorders) | 4 | 4
Itching (Skin and subcutaneous tissue disorders) | 6 | 5
Sleepiness (General disorders) | 7 | 3
Slow thinking (Nervous system disorders) | 3 | 3
Abnormal vision (Eye disorders) | 5 | 1
Eye pain (Eye disorders) | 3 | 4
Confusion (Nervous system disorders) | 4 | 6
Language problems (Nervous system disorders) | 4 | 3
Depression (Psychiatric disorders) | 3 | 3
Suicidal thoughts and actions (Psychiatric disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No